CLINICAL TRIAL: NCT06585202
Title: A Phase 2a Open-label Study to Investigate the Safety, Tolerability, Pharmacokinetics, Efficacy, and Pharmacodynamics of ATI-2138 Administered Over 12 Weeks in Participants With Moderate to Severe Atopic Dermatitis
Brief Title: Study of ATI-2138 in Adult Participants With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-2138-AD-201
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2024-11

CONDITIONS: Atopic Dermatitis
Keywords: Eczema; Dermatitis; Dermatitis, Atopic; Skin Diseases, Eczematous; Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Eczema; Dermatitis; Skin Diseases, Eczematous; Skin Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- ATI-2138 (Experimental): ATI-2138 oral tablets BID
  Interventions: Drug: ATI-2138

INTERVENTIONS:
Drug: ATI-2138 — ATI-2138 Oral Tablets BID

SUMMARY:
This is a Phase 2 open label study of ATI-2138 in participants with moderate to severe atopic dermatitis.

DETAILED DESCRIPTION:
This open-label, single-arm study of ATI-2138 in moderate to severe AD participants between the ages of 18 and 60 years (inclusive) will investigate the safety, tolerability, pharmacokinetics, efficacy and pharmacodynamics of ATI-2138 administered over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign the IRB approved ICF/assent prior to administration of study-related procedures.
* Male patients or non-pregnant, non-nursing female patients 18 to 60 years old, inclusive, at the time of informed consent/assent.
* Have at least a 1-year history of moderate or severe AD prior to the Screening Visit, and no significant AD flares for the 4 weeks prior to the Screening Visit as determined by the Investigator upon review of participant medical history.

Exclusion Criteria:

* Any prior exposure to systemic (oral) JAK inhibitors or TYK inhibitors at any time prior to Screening.
* Unstable course of AD (spontaneously improving or rapidly deteriorating) based on the patient history or as determined by the investigator during the Screening Period.
* Refractory AD (ie, AD that required frequent hospitalizations and/or frequent intravenous treatment for skin infections within the year before the Screening Visit).
* Concomitant skin disease or clinically infected AD or presence of other skin disease in the area to be dosed that may interfere with study assessments.
* Female patients who are pregnant, nursing, or planning to become pregnant during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | From baseline up to two weeks after treatment (Day 98)

SECONDARY OUTCOMES:
Change from baseline Eczema Area and Severity Index (EASI) Over Time | Up to Week 12
Proportions of participants who achieve at least 50%, 75%, and 90% improvement in EASI Over Time | Up to Week 12
Proportion of participants achieving Investigator's Global Assessment-Treatment Success Over Time | Up to Week 12
Change in IGA score over time | Up to Week 12
Change from baseline in AD Body Surface Area (BSA) over time | Up to week 12
Change from baseline in Peak Pruritus Numerical Rating Scale (PP-NRS) over time | Up to Week 12
ATI-2138 trough concentration ng/mL | Day 1 to Week 12
ATI-2138 peak concentration (Cmax) ng/mL | Day 1 to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Aggarwal, MD, Study Director — Aclaris Therapeutics, Inc.
Locations (6):
- United States (6):
  - Aclaris Investigational Site, Birmingham, Alabama
  - Aclaris Investigational Site, Encino, California
  - Aclaris Investigational Site, San Diego, California
  - Aclaris Investigational Site, Plainfield, Indiana
  - Aclaris Investigational Site, Austin, Texas
  - Aclaris Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No